CLINICAL TRIAL: NCT04455919
Title: Impact of Yoga on Quality of Life in Patients With Chronic Chikungunya: A Randomized Controlled Study
Brief Title: Yoga for Chronic Chikungunya
Acronym: YOCHIK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: covid health crisis
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PAP/RI2/2019_05; 2019-A01632-55 (Other: ANSM)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-07

CONDITIONS: Chikungunya Virus Infection
Keywords: chikungunya virus; yoga; chronic chikungunya
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: randomized wait-list controlled design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga (Experimental): Yoga classes once a week for eight weeks
  Interventions: Other: Yoga group
- Wait-list control (Other): The delayed intervention group was to benefit from the intervention after week 8.
  Interventions: Other: Wait-list group

INTERVENTIONS:
Other: Wait-list group — The wait-list group benefit from a 8-week yoga program after the interventional group
  Arms: Wait-list control
Other: Yoga group — During 8 weeks, the intervention group attended weekly yoga sessions and had to practice poses at home
  Arms: Yoga

SUMMARY:
The purpose of this study is to assess the benefits of a 8-week yoga program on quality of life in patients suffering from chronic chikungunya.

Studies have already shown the effectiveness of yoga practice on various arthralgia's, on the reduction of inflammatory reactions, on psychological disorders/sleep disorders and on quality of life. Considering quality of life as a global experience of balance between physical and mental wellbeing, the hypothesis was that the practice of yoga would globally improve the quality of life of patients with chronic chikungunya.

DETAILED DESCRIPTION:
The chikungunya virus (CHIKV) is an arbovirus passed to humans by Aedes mosquitoes. Since its description in 1952, CHIKV has caused millions of human infections in Africa, the Indian Ocean islands, Asia, Europe and America (1). In total, since 2013, the epidemic has affected more than 2 million people in the Americas. In Guadeloupe, the emergence of chikungunya cases began in 2013. CHINKV was declared an epidemic in 2014 with an estimated 20,000 infected patients.Human infection with CHIKV is characterized by a sudden onset of severe joint pains, high fever and rash. The infection is self-limited and acute symptoms usually disappear within one or two weeks. However, this polyarthralgia is recurrent in 30 to 40% of infected people and can persist for years. Chikungunya is considered chronic if the symptoms persist after three months. The chronic stage can last from a few months to several years. Chronic chikungunya usually manifests as joint pain and stiffness, polyarthralgia (including rheumatoid arthritis, flare-ups of spondylitis), and other general symptoms such as intermittent headaches, edema, and paresthesia. The consequences of chronic CHIKV can be severe, with patients becoming maladjusted to their lifestyle, feeling weakened and diminished. Depression and medical leaves are very frequent, with many cases of disability. Yoga is an ancestral Indian practice aiming to connect the "body" and the "soul", the "self" and "the other". Traditionally, it is a philosophical way of living, sometimes combined with the practice of physical exercises. In westernized countries, Yoga is usually considered as a physical practice or an alternative therapy, using various techniques of breathing, relaxation and poses to release tensions and decrease pain.

Studies have already shown the effectiveness of yoga practice on various arthralgia's, on the reduction of inflammatory reactions, on psychological disorders/sleep disorders and on quality of life. Considering quality of life as a global experience of balance between physical and mental wellbeing, the hypothesis was that the practice of yoga, by improving these different aspects, would globally improve the quality of life of patients with chronic chikungunya.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from chronic chikungunya, as documented by a positive chikungunya serology and the following symptoms: polyarthralgia and/or musculoskeletal disorder and/or morning stiffness.
* Patients had to be between 18 and 70 years old, and be
* patients affiliated to the French social insurance.

Exclusion Criteria:

* being pregnant;
* suffering from pre-existing rheumatic diseases before the Chikungunya infection;
* showing acute symptoms of a Chikungunya infection (documented serology);
* being unable to practice yoga poses ; having been recently treated with methotrexate or corticosteroids (less than 3 months ago);
* being under guardianship, trusteeship or legal protection,
* participating in another research study,
* showing severely impaired physical and/or psychological health, which in the opinion of the investigator, may affect the compliance of the study participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life - Short Form-36 (SF-36) | At baseline
  This scale measures eight health domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health) of quality of life for adults aged 18 and older. Using a scoring algorithm, the aggregated scores can provide two summary scores: the physical component summary (PCS) score and the mental component summary (MCS) score.
Health Related Quality of Life - Short Form-36 (SF-36) | after 8 weeks of intervention
  This scale measures eight health domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health) of quality of life for adults aged 18 and older. Using a scoring algorithm, the aggregated scores can provide two summary scores: the physical component summary (PCS) score and the mental component summary (MCS) score.
Health Related Quality of Life - Short Form-36 (SF-36) | after 18 weeks
  This scale measures eight health domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health) of quality of life for adults aged 18 and older. Using a scoring algorithm, the aggregated scores can provide two summary scores: the physical component summary (PCS) score and the mental component summary (MCS) score.

SECONDARY OUTCOMES:
nociceptive pain - Visual Analog Scale (VAS) | At baseline
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. They can also be asked to mark their maximum, minimum, and average pain. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no pain" anchor point.
nociceptive pain - Visual Analog Scale (VAS) | after 8 weeks of intervention
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. They can also be asked to mark their maximum, minimum, and average pain. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no pain" anchor point.
nociceptive pain - Visual Analog Scale (VAS) | after 18 weeks
  The Visual Analog Scale (VAS) is a 10 cm line with anchor statements on the left (no pain) and on the right (extreme pain). The patient is asked to mark their current pain level on the line. They can also be asked to mark their maximum, minimum, and average pain. The examiner scores the VAS by measuring the distance in either centimeters (0 to 10) or millimeters (0 to 100) from the "no pain" anchor point.
neuropathic pain- DN4 scale | At baseline
  The total score is calculated as the sum of the 10 items and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.
neuropathic pain- DN4 scale | after 8 weeks of intervention
  The total score is calculated as the sum of the 10 items and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.
neuropathic pain- DN4 scale | after 18 weeks
  The total score is calculated as the sum of the 10 items and the cut-off value for the diagnosis of neuropathic pain is a total score of 4/10.

CONTACTS AND LOCATIONS:
Locations (1):
- Mouffias' Medical Center in Guadeloupe., Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No